CLINICAL TRIAL: NCT06229340
Title: New Therapeutic Approaches for Tumors With RAS Gene Mutations
Brief Title: Leflunomide or Combination of MEK Inhibitor and Hydroxychloroquine for Refractory Patients With RAS Mutations
Acronym: NТО-RAS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Principal Investigator, Baboshkina Liliya Sergeevna, Oncologist, N.N. Petrov National Medical Research Center of Oncology
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LS01
Record Dates: First submitted 2023-12-21; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: RAS Mutation; Ras (Kras or Nras) Gene Mutation; Colorectal Cancer Recurrent; Pancreas Cancer; Lung Cancer; Melanoma; Refractory Cancer
Keywords: RAS Mutation; Ras (Kras or Nras) Gene Mutation; Colorectal Cancer; Pancreas Cancer; Melanoma; Lung Cancer; Refractory Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Lung Neoplasms; Melanoma; Neoplasms; Colorectal Neoplasms | interventions — Leflunomide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Leflunomide
  Interventions: Drug: Leflunomide
- Group 2 (Experimental): Combination of MEK Inhibitor and Hydroxychloroquine ( Plaquenil)
  Interventions: Drug: The combination of MEK inhibitor + hydroxychloroquine( plaquenil) ± bevacizumab
- historical control group (No Intervention): standard therapy

INTERVENTIONS:
Drug: Leflunomide — 100 mg daily for 3 days at the loading dose, then 20 mg daily at the standard dose.
  Arms: Group 1
Drug: The combination of MEK inhibitor + hydroxychloroquine( plaquenil) ± bevacizumab — Use of one of the possible MEK-inhibitor options:
  Trametinib 2 mg once daily orally; Cobimetinib 60 mg on days 1-21, break 7 days, cycle 28 days orally; Binimetinib 45 mg 2 times a day daily orally. + Hydroxychloroquine 600 mg 2 times a day daily orally.
  ± Bevacizumab 7.5 mg/m² every 3 weeks intravenously.
  Arms: Group 2

SUMMARY:
There is a huge variety of nucleotide substitutions that activate RAS. The search for new "universal" drugs for the RAS pathway that either interfere with RAS upregulation upstream in the signaling pathway or offset the consequences of RAS activation is important for improving therapeutic outcomes for patients with refractory malignancies.

The use of leflunomide or the combination of MEK inhibitor + hydroxychloroquine ± bevacizumab is promising for patients with mutations in RAS cascade genes who have failed all existing treatment standards.

DETAILED DESCRIPTION:
Mutations in the RAS gene are a common cause for the development of many tumors.

It is of practical interest to study the potential efficacy of several drugs registered for the treatment of other diseases, which may also be able to affect various parts of the RAS pathway.

Leflunomide, with its active metabolite , inhibits the enzyme dihydroorotate dehydrogenase (DHODH). DHODH plays an essential role in the biosynthesis of pyrimidine, which is particularly important for the growth of RAS mutant cells.

Tumors with KRAS, NRAS, and HRAS mutations are characterized by increased MEK kinase activity. The combination of MEK inhibitor + hydroxychloroquine ± bevacizumab is able to affect MEK kinase activity by direct inhibition as well as regulation of autophagy, which is controlled in this case by the antimalarial drug hydroxychloroquine.

The use of bevacizumab is appropriate because there is evidence of its efficacy in the treatment of patients with colorectal cancer, including colorectal cancer with mutations in the KRAS gene.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to provide informed consent and sign approved consent forms to participate in the study.
2. Patient age is at least 18 years old.
3. Performance status Eastern Cooperative Oncology Group (ECOG) 0-2.
4. Histologically confirmed metastatic metastatic disease stage 4.
5. Must have documented RAS (KRAS, HRAS, NRAS) mutation identified within the last 5 years by a local test on tumor tissue.
6. More than 2 lines of standard drug antitumor therapy in the anamnesis.
7. Must have disease progression as defined by RECIST version 1.1 criteria
8. Appropriate hematologic and liver function:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (1500/μL)
   * Lymphocyte count ≥ 0.5 x 109/L (500/μL)
   * Platelet count ≥ 100 x 109/L (100,000/μL) without transfusion
   * Hemoglobin ≥ 90 g/L without transfusion.
   * Creatinine clearance ≥ 40 mL/min
   * Serum albumin ≥ 25 g/L (2.5 g/dL)
   * Serum bilirubin ≤ 1.5 x HGH, with the following exception:
   * Patients with known Gilbert's disease or liver metastases: serum bilirubin level ≤ 3 x IUH
   * AST, ALT, and alkaline phosphate ≤ 2.5 x HGN;

10. For women of childbearing potential: consent to abstinence (abstain from heterosexual intercourse) or use at least two forms of effective contraception with an ineffectiveness rate < 1% per year during treatment.

11. Patients with asymptomatic new or advanced brain metastases (active brain metastases) are eligible to participate if the treating physician determines that localized treatment is not required.

Exclusion Criteria:

1. Age over 85 years.
2. Рresence of acute or active chronic infections.
3. Impaired renal and hepatic function; - left ventricular ejection fraction (LVEF) < 45%
4. Known history of acute or chronic hepatitis B or C due to known potential hepatotoxicity of leflunomide.
5. History of allergic reactions associated with compounds similar in chemical or biological composition to leflunomide or teriflunomide or other drugs in the combination.
6. Uncontrolled intercurrent disease, including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmias, or mental illness/social situations that limit study compliance.
7. Patients should not be pregnant or breastfeeding due to the potential for teratogenic effects and side effects of planned chemotherapeutic regimens.
8. History of retinal disease (retinal tear, exudate, hemorrhage) or retinal vein occlusion, central serous retinopathy or retinal pigment epithelium detachment, or current risk factors for ROS (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes).

Exit criteria:

1. Refusal to continue participation in the study.
2. Intolerable toxicity.
3. Progression according to RECIST 1.1 and IRECIST criteria or clinically significant (in the opinion of the physician) progression requiring a change in anticancer treatment.
4. Non-compliance with IND procedures.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | at the end of 2 cycles of treatment (each cycle is 28 days)
  Objective response rate was assigned for a subject if the subject displayed either complete response (CR) or partial response (PR) per RECIST version 1.1

SECONDARY OUTCOMES:
Assessment of patients' quality of life | at the end of 2 cycles of treatment (each cycle is 28 days)
  European Organization for the Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life (QoL) in cancer participants. It consisted of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, role, cognitive, emotional, social), and 9 symptom scales/items (Fatigue, nausea and vomiting, pain, dyspnoea, sleep disturbance, appetite loss, constipation, diarrhea, financial impact. The EORTC QLQ-C30 GHS/QoL score ranges from 0 to 100; High score indicates better GHS/QoL. Score 0 represents: very poor physical condition and QoL. Score 100 represents: excellent overall physical condition and QoL.
Progression-free survival (PFS) | at the end of 2 cycles of treatment (each cycle is 28 days)
  Progression-free survival was defined as the time from start treatment to subsequent confirmed progression per RECIST version 1.1, or death (whichever occurred first), measured in weeks and months. For PFS assessment clinical progression (i.e., treatment discontinuation due to progression of disease) was also considered as an event.
Overall survival | up to 3 years
  Overall survival was defined as the time from start treatment to subsequent death, measured in weeks and months.

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Imyanitov, Study Director — N.N. Petrov NMRC of Oncology
Locations (1):
- Department of Tumor Growth Biology, N.N. Petrov Institute of Oncology, Saint Petersburg, Russian Federation, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No